CLINICAL TRIAL: NCT02677181
Title: Prospective Study of Combined ATG Regimen for Prophylaxis of aGVHD in Matched Sibling Donor PBSCT
Brief Title: Efficacy and Safety Study of ATG for Prophylaxis of aGVHD in Matched Sibling Donor PBSCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: 309th Hospital of Chinese People's Liberation Army (Other); Beijing Naval General Hospital (Other); Space Center Hospital, Peking University (Unknown)
Responsible Party: Principal Investigator, Daihong Liu, Head of Hematology departemnt in Chinese PLA General Hospital, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 81370666
Record Dates: First submitted 2015-12-01; First posted 2016-02-09 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: aGVHD
Keywords: ATG; Matched sibling donor; peripheral blood stem cell transplantation
MeSH Terms: interventions — Antilymphocyte Serum; Cyclosporins; Mycophenolic Acid; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATG combined regimen (Experimental): ATG combined regimen for prophylaxis of GVHD, includes ATG, MMF(Mycophenolate mofetil ),CsA (cyclosporin A) and MTX (methotrexate).
  All recipients in this arm received ATG, CsA, mycophenolate mofetil, and short-term methotrexate for GVHD prophylaxis. ATG (Thymoglobuline, rabbit) was used as 1.5 mg/kg/d on day -5 and 3.5 mg/kg/d on day -4. CsA (3 mg/kg, q12h, i.v.) was used from day -9, and the concentration was adjusted to 180-200 ng/mL. CsA was switched to oral administration when the patient's bowel function recovered. From day -9, 0.5 g of mycophenolate mofetil was administered orally from every 12 h, which was withdrawn on day +30. After graft infusion, MTX was given for all patients at 15 mg/m2 on day +1 and 10 mg/m2 on days +3, +6 and +11.
  Interventions: Drug: ATG; Drug: CsA; Drug: mycophenolate mofetil; Drug: Methotrexate
- no-ATG (Active Comparator): regimen for prophylaxis of GVHD without ATG. The regimen includes MMF,CsA and MTX.CsA (3 mg/kg, q12h, i.v.) was used from day -9, and the concentration was adjusted to 180-200 ng/mL. CsA was switched to oral administration when the patient's bowel function recovered. From day -9, 0.5 g of mycophenolate mofetil was administered orally from every 12 h, which was withdrawn on day +30. After graft infusion, MTX was given for all patients at 15 mg/m2 on day +1 and 10 mg/m2 on days +3, +6 and +11.
  Interventions: Drug: CsA; Drug: mycophenolate mofetil; Drug: Methotrexate

INTERVENTIONS:
Drug: ATG — rabbit ATG（Sanofi）
  Other Names: Thymoglobuline
  Arms: ATG combined regimen
Drug: CsA — cyclosporine (3 mg/kg, q12h, i.v.) was used from day -9, and the concentration was adjusted to 180-200 ng/mL. CsA was switched to oral administration when the patient's bowel function recovered.
  Other Names: Neoral/Sandimmun
Drug: mycophenolate mofetil — From day -9, 0.5 g of mycophenolate mofetil was administered orally from every 12 h, which was withdrawn on day +30 for MSD-PBSCT.
  Other Names: MMF（Novartis）
Drug: Methotrexate — short-term methotrexate
  Other Names: MTX(Pfizer)

SUMMARY:
The purpose of this study is to determine the efficacy and safety of combined ATG （antithymocyte globulin ） regimen for aGVHD(acute graft-versus-host disease ) prophylaxis in matched sibling donor peripheral blood stem cell transplantation (MSD-PBSCT).

DETAILED DESCRIPTION:
Transplantation with G-CSF （Granulocyte colony stimulating factor ）mobilized peripheral blood stem cell (PBSCT) has been a stable transplant setting with matched sibling donor transplantation. Unmanipulated haploidentical donor PBSCT (haplo-PBSCT) has been applied in patients with hematologic malignancies. In our previous cohort study, haplo-PBSCT was associated with lower incidence of severe acute GVHD and extensive chronic GVHD compared with matched sibling donor PBSCT (MSD-PBSCT). Haplo-PBSCT has the same GVHD prophylaxis regimen with MSD-PBSCT, except ATG. It suggested the potential advantage of ATG in prophylaxis of GVHD and improvement of long-term quality of life of the transplant recipients, which motivate us to observe the efficacy of combined ATG regimen for GVHD prophylaxis in MSD-PBSCT.

ELIGIBILITY:
Inclusion Criteria:

1. acute myeloid leukemia (AML) in CR1 (complete remission 1) or CR2 (complete remission 2) phase regardless of cytogenetics;
2. CML CP(chronic myelogenous leukemia , chronic phase); NHL (non-Hodgkin's lymphoma )
3. MDS-RAEB(myelodysplastic syndrome -refractory anemia with excess blasts ).
4. All patients should aged 40 to 70 years
5. Have matched sibling donor.
6. Patients without any uncontrolled infections or without severe pulmonary, renal, hepatic or cardiac diseases .

Exclusion Criteria:

1. Patients aged less than 40 years old ;
2. Patients with any uncontrolled infections or with severe pulmonary, renal, hepatic or cardiac diseases;
3. AML patients with t (15;17);

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with cGVHD as assessed by chronic graft versus host disease grading criteria (refer to NIH criteria) | three years
  Chronic graft versus host disease grading criteria (refer to NIH criteria)

SECONDARY OUTCOMES:
all cause mortality | two years
Number of participants relapse as assessed by NCCN (National Comprehensive Cancer Network )criteria | two years
DFS(disease-free survival ) | two years
  disease-free survival
TRM(treatment-related mortality ) | two years
  treatment-related mortality
Number of participants with aGVHD as assessed by acute graft versus host disease grading criteria (refer to Glucksberg criteria) | three months

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Doctor, Study Director — Chinese PLA General Hospital
Locations (1):
- Liping Dou, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armand P, Kim HT, Zhang MJ, Perez WS, Dal Cin PS, Klumpp TR, Waller EK, Litzow MR, Liesveld JL, Lazarus HM, Artz AS, Gupta V, Savani BN, McCarthy PL, Cahn JY, Schouten HC, Finke J, Ball ED, Aljurf MD, Cutler CS, Rowe JM, Antin JH, Isola LM, Di Bartolomeo P, Camitta BM, Miller AM, Cairo MS, Stockerl-Goldstein K, Sierra J, Savoie ML, Halter J, Stiff PJ, Nabhan C, Jakubowski AA, Bunjes DW, Petersdorf EW, Devine SM, Maziarz RT, Bornhauser M, Lewis VA, Marks DI, Bredeson CN, Soiffer RJ, Weisdorf DJ. Classifying cytogenetics in patients with acute myelogenous leukemia in complete remission undergoing allogeneic transplantation: a Center for International Blood and Marrow Transplant Research study. Biol Blood Marrow Transplant. 2012 Feb;18(2):280-8. doi: 10.1016/j.bbmt.2011.07.024. Epub 2011 Jul 31. PMID 21810400
- [Background] Rezvani AR, Storb RF. Prevention of graft-vs.-host disease. Expert Opin Pharmacother. 2012 Aug;13(12):1737-50. doi: 10.1517/14656566.2012.703652. Epub 2012 Jul 7. PMID 22770714
- [Background] Storb R, Deeg HJ, Whitehead J, Appelbaum F, Beatty P, Bensinger W, Buckner CD, Clift R, Doney K, Farewell V, et al. Methotrexate and cyclosporine compared with cyclosporine alone for prophylaxis of acute graft versus host disease after marrow transplantation for leukemia. N Engl J Med. 1986 Mar 20;314(12):729-35. doi: 10.1056/NEJM198603203141201. PMID 3513012
- [Background] Finke J, Bethge WA, Schmoor C, Ottinger HD, Stelljes M, Zander AR, Volin L, Ruutu T, Heim DA, Schwerdtfeger R, Kolbe K, Mayer J, Maertens JA, Linkesch W, Holler E, Koza V, Bornhauser M, Einsele H, Kolb HJ, Bertz H, Egger M, Grishina O, Socie G; ATG-Fresenius Trial Group. Standard graft-versus-host disease prophylaxis with or without anti-T-cell globulin in haematopoietic cell transplantation from matched unrelated donors: a randomised, open-label, multicentre phase 3 trial. Lancet Oncol. 2009 Sep;10(9):855-64. doi: 10.1016/S1470-2045(09)70225-6. Epub 2009 Aug 18. PMID 19695955
- [Background] Wang Y, Fu HX, Liu DH, Xu LP, Zhang XH, Chang YJ, Chen YH, Wang FR, Sun YQ, Tang FF, Liu KY, Huang XJ. Influence of two different doses of antithymocyte globulin in patients with standard-risk disease following haploidentical transplantation: a randomized trial. Bone Marrow Transplant. 2014 Mar;49(3):426-33. doi: 10.1038/bmt.2013.191. Epub 2013 Dec 2. PMID 24292519
- [Background] Hamadani M, Blum W, Phillips G, Elder P, Andritsos L, Hofmeister C, O'Donnell L, Klisovic R, Penza S, Garzon R, Krugh D, Lin T, Bechtel T, Benson DM, Byrd JC, Marcucci G, Devine SM. Improved nonrelapse mortality and infection rate with lower dose of antithymocyte globulin in patients undergoing reduced-intensity conditioning allogeneic transplantation for hematologic malignancies. Biol Blood Marrow Transplant. 2009 Nov;15(11):1422-30. doi: 10.1016/j.bbmt.2009.07.006. Epub 2009 Sep 1. PMID 19822302
- [Background] Storek J, Mohty M, Boelens JJ. Rabbit anti-T cell globulin in allogeneic hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2015 Jun;21(6):959-70. doi: 10.1016/j.bbmt.2014.11.676. Epub 2014 Dec 5. PMID 25482864
- [Derived] Chakupurakal G, Freudenberger P, Skoetz N, Ahr H, Theurich S. Polyclonal anti-thymocyte globulins for the prophylaxis of graft-versus-host disease after allogeneic stem cell or bone marrow transplantation in adults. Cochrane Database Syst Rev. 2023 Jun 21;6(6):CD009159. doi: 10.1002/14651858.CD009159.pub3. PMID 37341189
- [Derived] Dou L, Wang L, Li X, Liu Y, Li F, Wang L, Gao X, Huang W, Wang S, Gao C, Yu L, Liu D. Role of antithymocyte globulin in matched sibling donor peripheral blood stem cell transplantation for hematologic malignancies. Medicine (Baltimore). 2021 Feb 26;100(8):e24725. doi: 10.1097/MD.0000000000024725. PMID 33663084